CLINICAL TRIAL: NCT03976947
Title: Impact of Lung Recruitment Maneuvers on Driving Pressure in Cardiac Surgery (IMPREMO): Before - After Trial
Brief Title: Impact of Lung Recruitment Maneuvers on Driving Pressure in Cardiac Surgery
Acronym: IMPREMO
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 17-023
Record Dates: First submitted 2017-04-14; First posted 2019-06-06 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2019-06

CONDITIONS: Respiration, Artificial; Lung Diseases; Atelectasis; Cardiac Surgical Procedures; Anesthesia, General
Keywords: Driving pressure; Postoperative pulmonary complications
MeSH Terms: conditions — Respiratory Aspiration; Lung Diseases; Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Before group: The "before" group is the control group. We collect retrospective data in consecutive patients operated before the implementation of lung recruitment maneuvers protocol
- After group: We collect data in consecutive patients operated after the implementation of lung recruitment maneuvers protocol. This lung recruitment maneuvers will be realised along the surgery, (After tracheal intubation, per-CPB, post-CPB). Each recruitment maneuver consisted of applying a continuous positive airway pressure of 30 cm of water for 30 seconds

SUMMARY:
In anesthesia the incidence of postoperative pulmonary complications is frequent, especially in cardiac surgery where the incidence can reach 10%. Respiratory morbidity in cardiac surgery is favored by multiple factors and is higher compared to anesthesia in "general" surgery. The prevention of these complications is a major challenge in the management of patients.

Influence of driving pressure level on respiratory morbidity was first demonstrated in management of acute respiratory distress syndrome (ARDS) in resuscitation.

More recently, this notion has been introduced in anesthesia, with a correlation between increase driving pressure level and increase of post-operative respiratory complications.

A method should reduce these levels of driving pressure: performing lung recruitment maneuvers. This technique has been successfully tested in abdominal surgery in particular in a study published by Futier et al.. They systematized and standardized lung recruitment maneuvers and showed a decrease of postoperative pulmonary complications in abdominal surgery.

Thus, the realization of lung recruitment maneuvers, already used at the discretion of the practitioner, is now recommended by several teams of experts. The investigators propose in this "before-after" trial to evaluate variation in driving pressure due to systematic use of lung recruitment maneuvers, observed in patients operated in elective or urgent surgery. The secondary objective is to evaluate their impact on postoperative pulmonary complications.

DETAILED DESCRIPTION:
This is a retrospective, before / after, monocentric trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving elective or urgent cardiac surgery with cardiopulmonary bypass

Exclusion Criteria:

* Emergency or salvage surgery
* Patient under guardianship
* Pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients receiving cardiac surgery with cardiopulmonary bypass
Sampling Method: Probability Sample
Enrollment: 217 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Driving pressure variation due to lung recruitment maneuvers | 1 day
  cmH2O

SECONDARY OUTCOMES:
Incidence of postoperative pulmonary complications | baseline
  percentage

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Brunet, MD, Principal Investigator — University Hospital of Caen
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neto AS, Hemmes SN, Barbas CS, Beiderlinden M, Fernandez-Bustamante A, Futier E, Gajic O, El-Tahan MR, Ghamdi AA, Gunay E, Jaber S, Kokulu S, Kozian A, Licker M, Lin WQ, Maslow AD, Memtsoudis SG, Reis Miranda D, Moine P, Ng T, Paparella D, Ranieri VM, Scavonetto F, Schilling T, Selmo G, Severgnini P, Sprung J, Sundar S, Talmor D, Treschan T, Unzueta C, Weingarten TN, Wolthuis EK, Wrigge H, Amato MB, Costa EL, de Abreu MG, Pelosi P, Schultz MJ; PROVE Network Investigators. Association between driving pressure and development of postoperative pulmonary complications in patients undergoing mechanical ventilation for general anaesthesia: a meta-analysis of individual patient data. Lancet Respir Med. 2016 Apr;4(4):272-80. doi: 10.1016/S2213-2600(16)00057-6. Epub 2016 Mar 4. PMID 26947624
- [Background] Futier E, Constantin JM, Paugam-Burtz C, Pascal J, Eurin M, Neuschwander A, Marret E, Beaussier M, Gutton C, Lefrant JY, Allaouchiche B, Verzilli D, Leone M, De Jong A, Bazin JE, Pereira B, Jaber S; IMPROVE Study Group. A trial of intraoperative low-tidal-volume ventilation in abdominal surgery. N Engl J Med. 2013 Aug 1;369(5):428-37. doi: 10.1056/NEJMoa1301082. PMID 23902482